CLINICAL TRIAL: NCT04302623
Title: Meditation and Yoga for Irritable Bowel Syndrome Study
Brief Title: Meditation and Yoga for Irritable Bowel Syndrome
Acronym: MY-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Maitreyi Raman, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REB20-0084
Record Dates: First submitted 2020-02-29; First posted 2020-03-10 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Yoga; Meditation; Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Yoga; Meditation; eHealth; Quality of Life
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online yoga program (Experimental): An 8-week online live facilitator-led yoga program.
  Interventions: Behavioral: Yoga
- Control (Experimental): Advice only group.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Upa Yoga program consisting of physical postures, breathing techniques, chanting, and meditation.

SUMMARY:
Study Aim: This study will explore the feasibility and effectiveness of a yoga program for patients with IBS.

Methods: A superiority RCT with 30 participants per group. Adult patients with IBS fluent in English who do not have major physical impairments or cognitive, psychological, or psychiatric disorder will be recruited and randomly using the REDCap randomization module to either a yoga intervention delivered (a) a yoga intervention delivered online led by a yoga facilitator or (b) a advice only control group. The 8-week Hatha Yoga intervention consists of Yoga Namaskar, Nadi Shuddhi (alternate nostril breathing), mantra chanting, and breath watching.

Group 1: Yoga program. Participants will be asked to practice the yoga program daily at home and will be given access to the yoga videos hosted on the University of Calgary study website, as well as written program instructions, and frequently answered questions. A brief description of the video content will be provided to inform the participant of its content and length. Additional website content will include study information, study schedule, and contact information, as well as a pre-recorded educational session. In addition to the daily program describe above, the facilitator-led intervention will be delivered online by a certified yoga facilitator using the Microsoft Teams platform. Participants in group of 3 to 5 will be collated to enhance effectiveness of the study processes. Our team has experience with this approach, as this strategy is currently used with previous yoga study. Yoga classes will be held once per week for 8 weeks, with the first session lasting approximately 1.5 hours and subsequent sessions up to 60 minutes. The total allocated time for the introductory session will include the class set-up, introductions, educational material (please see below), overview of practices, teaching of practices, practice corrections/enhancements, modifications, and practice expectations. Each follow-up class will include review from the previous week, questions and answers, individual corrections and/or modifications. For individual corrections, the yoga facilitator will ask the participant to do the practices and receive corrections, if needed.

Group 2. Advice-only control group. This group will receive general education on IBS, the mind and gut connection, and the role of mind-body therapies in the management of IBS.

Effectiveness outcomes will be assessed at baseline and 8 weeks. The primary effectiveness outcome will be the severity of IBS symptoms, and secondary effectiveness outcomes include microbiome analysis, quality of life, anxiety and depression symptoms, perceived stress, fatigue, and severity of somatic symptoms. Microbiome composition will be measured using shotgun metagenomic sequencing. Microbiome sequences will be analyzed for alpha diversity, beta diversity, species composition, functional composition and biomarker discovery. To determine the feasibility of each intervention, recruitment and attrition rates, adherence, program preferences and satisfaction, and adverse event outcomes will be evaluated.

DETAILED DESCRIPTION:
Study Aim. This study will explore the feasibility and effectiveness of a yoga program for patients with IBS. Objective. Examine the feasibility and effectiveness of an 8-week online live facilitator-led yoga program compared to a wait-list control. Hypothesis. Yoga delivered online live by a facilitator will have the superior effectiveness in reducing IBS symptoms compared to advice only control group after 8 weeks.

Background

IBS is a highly prevalent disorder affecting 12% of Canadians. One in five individuals with IBS has one or more psychiatric disorder, and 50% have at least one comorbid somatic symptom. Frequently used therapies are targeted toward symptom reduction with modest benefits, whereas treatments with greater therapeutic effect may be associated with side effects. This leaves many patients dissatisfied with their symptom management, resulting in half of patients using alternative therapies. The underlying cause of IBS is likely multifactorial and the interplay of the brain-gut axis in the pathophysiology of IBS has been well established. An altered stress response, arising through either psychological and/or physiological mechanisms is hypothesized to be involved in the impairment of the signalling between the brain and the gut. This demonstrates a connection between gut function, stress, and psychological processes. Therefore, therapies that focus on mind-body interactions and stress reduction, may be useful adjunctive treatments for IBS.

Yoga is a traditional "mind-body-breath" discipline that includes yogic postures, structured breathing, and meditation. Several potential mechanisms for the effectiveness of yoga that have applicability to IBS have been proposed, including reducing the upregulated sympathetic activity and increasing the parasympathetic response. The investigator's recent review of the literature has identified four randomized controlled trials that examined traditional yoga practice as therapy for adult IBS patients. All trials found yoga as more effective compared to pharmacological treatment, and equally effective as dietary interventions or moderate-intensity walking. Both physical (IBS symptom severity, gastric motility, autonomic and somatic symptom scores, physical functioning) and mental (depression, anxiety, GI-specific anxiety, and QOL) improvements were seen. The current literature supports that yoga is effective, safe and it may target multiple mechanisms involved in the treatment of IBS symptoms as previously described. Although yoga is effective in managing IBS symptoms, further research is needed to determine the feasibility and effectiveness of yoga as a therapeutic option in clinical practice for patients with IBS, while also examining delivery strategies (face-to-face vs. online) to more optimally understand how to sequence therapeutic interventions and whether this improves initiation and adherence to the intervention.

Research Methods

Study Design. Superiority trial.

Recruitment. Potential participants will be identified through several avenues, including:

1. Gastroenterologists will screen IBS patients using the study eligibility criteria and following the patient's verbal consent, will share the patient's contact information with the study coordinator. Patients have previously given verbal permission at the clinic to their gastroenterologist to be asked to participate in research studies.
2. Self-referral through poster advertising in the GI clinics at Foothills and South Health Campus. In addition, the study will be advertised on the Faculty of Medicine TVs on the Foothills campus.
3. IMAGINE (Inflammation, Microbiome and Alimentation Gastro-intestinal and Neuropsychiatric Effects) cohort study at the University of Calgary: The IMAGINE study will send an initial email to all its IBS patients who have consented to be contacted for future studies. This email will explain the current study and connect interested participants with the study coordinator.
4. Self-referral through the Primary Care Networks (PCNs) in Calgary. Primary care physicians and/or dieticians (depending on the PCN clinic) will inform their IBS patients of the study and provide the patient with a brochure.
5. Through the use of a privately owned Facebook group called 'Low FODMAP Canadians', a group managed by two Canadian dieticians Lauren Renlund, MPH, RD and Audrey Inouye, RD. This group has over 2.1K members who have IBS.
6. Participants who indicated interest in this study in a previous survey (REB19-1456) and have given their consent to be contacted.

Screening. Consented participants will complete a mental health evaluation using the Patient Health Questionnaire-9 (PHQ-9). Individuals who score 20 points or higher on the PHQ-9 indicating sever depression will not be eligible to participate.

Intervention. Participants will be assigned randomly using the REDCap randomization module to either (a) a yoga intervention delivered online led by a yoga facilitator or (b) a advice only control group. The intervention group will receive a yoga program described below called Upa Yoga, including yoga Namaskar, Nadi Shuddi (alternate nostril breathing), mantra meditation, and breath watching. The intervention was developed in keeping with the ancient principles of Hatha Yoga and delivered by a trained yoga facilitator from the Isha Yoga Institute of Inner Sciences.

* Yoga Namaskar activates the lumbar region of the spine and strengthens the core muscles. This set of practices involves a series of 7 steps including stretching, squatting and structured breathing sequences which will take 10 minutes to complete.
* Nadi Shuddhi or alternate nostril breathing helps to bring balance between activity and emotion. Participants will sit in a cross-legged posture with the spine comfortably erect, eyes closed with the left hand laced in the middle of the lap, palm facing upwards, and the ring and index finger will be used to block one nostril while inhaling and exhaling through the other. This practice takes a minimum of 5 minutes to complete.
* Mantra Meditation. In the yogic culture, the entire existence is seen as a web of sounds or vibrations, for which the root sounds are "Aa, Oo, and Mm". These three sounds are referred to as universal sounds. This mantra, Aum, facilitates energy flow, and through vibratory mechanisms, has been demonstrated to create peace and harmony. This will be practiced for 3 minutes.
* Breath Watching. The science of breath watching in the yogic literature, employs the following principle: a certain thought, emotion or change in the physical body might change the breath flow. Similarly, the converse of principle is true, in that breathing in a structured manner can be used as a tool to bring positive changes to the practioners' mind, body and emotions. The practioners will assume a specific cross-legged physical posture, and practice breath watching as guided by the yoga instructor for 3-5-minutes.

Group 1: Yoga program. Participants will be asked to practice the yoga program daily at home and will be given access to the yoga videos hosted on the University of Calgary study website, as well as written program instructions, and frequently answered questions (Appendix A). A brief description of the video content will be provided to inform the participant of its content and length. Additional website content will include study information, study schedule, and contact information, as well as a pre-recorded educational session.

In addition to the daily program describe above, the facilitator-led intervention will be delivered online by a certified yoga facilitator using the Microsoft Teams platform. Participants in group of 3 to 5 will be collated to enhance effectiveness of the study processes. Our team has experience with this approach, as this strategy is currently used with previous yoga study. Yoga classes will be held once per week for 8 weeks, with the first session lasting approximately 1.5 hours and subsequent sessions up to 60 minutes. The total allocated time for the introductory session will include the class set-up, introductions, educational material (please see below), overview of practices, teaching of practices, practice corrections/enhancements, modifications, and practice expectations. Each follow-up class will include review from the previous week, questions and answers, individual corrections and/or modifications. For individual corrections, the yoga facilitator will ask the participant to do the practices and receive corrections, if needed.

Group 2. Advice-only control group. This group will receive general education on IBS, the mind and gut connection, and the role of mind-body therapies in the management of IBS.

Educational Material. The intervention group will receive educational material consisting of information on IBS, why yoga may improve IBS symptoms and quality of life, and self-compassion (Appendix B) during their first online session delivered by the study coordinator and yoga facilitator.

The study coordinator will orient each participant to the study, guide group 1 participants through expectations of the class, answer any study-related questions for the duration of the study. A study schedule will be provided to participants at the start of the study (Appendix C). The yoga facilitator will act as a point of contact to answer any questions related to the yoga program.

Practice Modifications. Intervention participants will receive modifications from the yoga facilitator for common challenges encountered by yoga practitioners to support optimal practices. Modifications will be provided in the online sessions.

Long-term follow-up. Yoga practice maintenance will be evaluated long-term. Intervention participants will be asked to report the average frequency (i.e., days per month) and length (i.e., minutes) of their yoga practices over the last 7 days at 6 months post intervention.

Feasibility outcomes. To determine the feasibility of each intervention, the following outcomes will be evaluated: recruitment and attrition rates, adherence, and satisfaction, and adverse event outcomes.

Sample size. 25 participants per group (mean difference of at least 83 points on the IBS-Symptom Severity Scale; ⍺=0.05, β=0.80, SD=103.8, ∆=83)35. Assuming a 20% attrition rate, we will aim to recruit 30 individuals per group.

Data Analysis. Descriptive analysis will summarize participant characteristics and feasibility outcomes. Independent sample t-tests will examine baseline differences between groups and chi-squared tests will examine proportion differences. Repeated measures ANOVA will examine the main effect of treatment condition and interactions of group assignment by time on effectiveness outcome measures. An alpha of 0.05 will be set a priori and used as a threshold for determining statistical significance. Analysis will be conducted using SPSS version 24.0.

For microbiome sequencing data quality control of raw FASTQ files will be performed, prior to ML analysis, to obtain high-quality non-host (HQNH) reads. Reads of sufficient quality will be mapped using MetaPhlAn2 and HUMAnN2 to obtain high-resolution taxonomic and functional abundance profiles that include read counts. Unsupervised learning strategy based on robust PCA will be used to explore the major variability in the data and to detect outliers. We will also perform KEGG annotations and functional diversity profiling and will use web-based tools to assign metagenomic results into different functional groups.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of IBS based on Rome IV criteria
* At least 18 years old
* Adequate understanding of English
* Ability to provide written informed consent
* No changes in IBS medication (including anti-depressants), diet, or physical activity levels for at least 8 weeks prior to starting the intervention

Exclusion Criteria:

* Major physical impairment that would prevent the individual from doing yoga
* Diagnosis of any major cognitive, psychological, or psychiatric disorder (diagnosed before or during the intervention) as identified by the treating physician/healthcare practitioner or screened by the study coordinator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
IBS-Symptom Severity Scale | Baseline and 8 weeks
  Scores range from 0 to 500 with higher scores indicating more severe symptoms. Symptom reduction of at least 50 points is considered clinically meaningful; however, the primary endpoint will be the proportion of participants in each group who demonstrate a symptom reduction of 83 points or more, based on the variables used in the sample size calculation.

SECONDARY OUTCOMES:
IBS-Quality of Life | Baseline and 8 weeks
  Scores range fro 34 to 170 with higher scores indicating better quality of life. An increment of at least 14 points from baseline will demonstrate efficacy.
Generalized Anxiety Disorder | Baseline and 8 weeks
  Scores range from 0 to 21. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety. A 5-point change is considered clinically significant.
Patient Health Questionnaire-9 (Depression) | Baseline and 8 weeks
  Scores range from 0 to 27. Scores of 5, 10, 15, and 20 represent cut points for mild, moderate, moderately severe and severe depression. A 5-point change is considered clinically significant.
Perceived Stress Scale | Baseline and 8 weeks
  Scores range from 0 to 44 with higher scores indicating more stress. A minimally clinical important change is at least 11 points.
Modified Fatigue Impact Scale-21 | Baseline and 8 weeks
  Scores range from 0 to 84, with higher scores indicating higher fatigue. A minimally clinically important difference is considered a change of at least 16 points on a 84-point scale.
Patient Health Questionnaire-15 (Somatic Symptoms) | Baseline and 8 weeks
  Scores range from 0 to 30. scores of 5, 10, and 15 represent cut points for low, medium, and high somatic symptom severity. Patient Health Questionnaire-15. A 5-point change is considered clinically significant.
COVID-19 Stress Scale | Baseline and 8 weeks
  COVID-19 related stress and anxiety will be measured using the 36-item CSS survey on five scales: (1) COVID danger and contamination fears, (2) COVID fears about economic consequences, (3) COVID xenophobia, (4) COVID compulsive checking and reassurance seeking, and (5) COVID traumatic stress symptoms.
Self-Compassion Scale-Short Form | Baseline and 8 weeks
  12-item self-reported scale measuring their self-compassion, including self-kindness, self-judgement, humanity, isolation, and mindfulness subscales. Subscale scores are computed by calculating the mean of subscale items responses. Participants will indicate how often they behave in the stated manner, using a scale from 1 (almost never) to 5 (almost always) for a total of 60 points with lower scores indicating more self-compassion
Recruitment rates | 8 weeks
  Recruitment rates will be calculated from the percentage of participants who complete the pre-screening, eligibility, and enrollment phases of the study.
Attrition rates | 8 weeks
  Calculated as the percentage of participants who complete all study measures. A retention rate of 70 percent will be deemed feasible (i.e., a drop-out rate of less than 30 percent from both groups combined).
Adherence to class attendance and home practice | 8 weeks
  Class attendance and home practice will be collected for 8 weeks. Total practice minutes will be added over the course of 8 weeks between class and home practice. Adherence will be defined as practicing daily yoga for at least 80 percent of days for 8 weeks (or minimum of 45 out of 56 days).
Program preferences | Baseline
  At the start of the study, participants will be asked if they have a preference on delivery modality (face-to-face or web-based). The relationship between program preference and adherence to the program will be examined.
Program satisfaction | 8 weeks
  Participants will complete a survey regarding overall satisfaction with their respective program, including satisfaction with website and video use and class instruction.
Adverse event outcomes | 8 weeks
  Participants will be asked to report to the study staff any adverse events experienced during the 8-week study period, regardless of their potential relationship to the intervention. Patients who report any events will be advised to consult their physician to assess the event and provide care as appropriate.
Intention to practice yoga | Baseline and 8 weeks
  Intention to practice yoga will be measured from 1 (very unlikely) to 7 (very likely) with "I intend to do yoga daily for 30-40 minutes for the next eight weeks". Values 1-3 will indicate low intention, 4=neutral, and values 5-7 will indicate high intention.

CONTACTS AND LOCATIONS:
Overall Officials: Maitreyi Raman, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available upon reasonable request from the study principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be shared when the manuscript has been published and the graduate student leading this study has defended their thesis (approximately Fall 2022). The data will be available for six months.
Access Criteria: Future collaboration (e.g., systematic review/meta-analysis).

REFERENCES:
- [Derived] D'Silva A, Marshall DA, Vallance JK, Nasser Y, Rajagopalan V, Szostakiwskyj JH, Raman M. Meditation and Yoga for Irritable Bowel Syndrome: A Randomized Clinical Trial. Am J Gastroenterol. 2023 Feb 1;118(2):329-337. doi: 10.14309/ajg.0000000000002052. Epub 2022 Oct 11. PMID 36422517
- [Derived] D'Silva A, Marshall DA, Vallance J, Nasser Y, Rajagopalan V, MacKean G, Raman M. Meditation and yoga for irritable bowel syndrome: study protocol for a randomised clinical trial (MY-IBS study). BMJ Open. 2022 May 26;12(5):e059604. doi: 10.1136/bmjopen-2021-059604. PMID 35618329